CLINICAL TRIAL: NCT02889094
Title: Multi-center Study Evaluating Persistence of Hepatitis B Virus Replication, Long-term Prognostic Indicators and Their Clinical Relevance in Patients Co-infected With the Human Immunodeficiency Virus and Chronic Hepatitis B
Brief Title: French HIV-HBV Cohort
Acronym: COVViB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Sidaction (Other)
Responsible Party: Sponsor
Other Study IDs: IMEA 49
Record Dates: First submitted 2016-08-25; First posted 2016-09-05 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis B; HIV; Liver Cirrhosis; End Stage Liver Disease
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be stored for quantification of biochemical parameters.
  Liver tissue (for individuals receiving liver biopsies) will be stored for quantification of intracellular HBV DNA replication.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV-HBV co-infected individuals: No interventions will be administered. Individuals will be undergoing routine care.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — Routine care recommended for patients co-infected with HIV and hepatitis B virus (per European Association for the Study of the Liver and European AIDS Clinical Society guidelines).

SUMMARY:
The overarching purpose of this study is to further understand the reasons for and clinical implications of persistent HBV infection in patients co-infected with HIV and HBV in the era of highly effective antiviral treatment against both viruses.

DETAILED DESCRIPTION:
The French HIV-HBV Cohort is an observational, non-interventional study including 308 HIV-infected patients with chronic HBV infection (HBsAg-positive serology >6 months) in seven clinical centers. Patients were recruited in 2002-2003 and followed prospectively every three to twelve months, during two phases, until 2010-2011. Extensive information on a variety of HIV- and HBV-related parameters were collected during these study visits.

This particular study aims to extend follow-up of the French HIV-HBV Cohort using a different type of design. Patients who completed at least one study phase of the French HIV-HBV Cohort are selected for participation. Patients continuing follow-up at a participating clinical center are asked to undergo their routine clinical visit, during which time medical data from the years since last cohort visit until their routine visit are extracted. For those who died, information from the years since last cohort visit until death will be collected.

The primary objective for this cohort extension is to further understand the reasons for and clinical implications of persistent HBV infection in patients co-infected with HIV and HBV in the era of highly effective antiviral treatment against both viruses.

The following secondary objectives are as follows:

* To establish the extent of persistent viremia (PV) of HBV, quantified either in serum or within the hepatocyte
* To understand whether this persistence effects clinically-relevant serological outcomes (i.e. HBeAg and HBsAg seroclearance and seroconversion along with HBsAg quantification) after prolonged follow-up
* To quantify the evolution of liver fibrosis using non-invasive methods and, in a small subset of patients, liver biopsies, while investigating the virological and immunological factors associated with its progression and regression
* To describe the causes of liver-related and non-liver-related morbidity and mortality and the direct effect of persistent HBV DNA replication on these outcomes

ELIGIBILITY:
Inclusion Criteria:

* HBsAg seropositivity for >6 months (at initial cohort inclusion)
* HIV-positive serology confirmed with Western blot (at initial cohort inclusion)
* Karnofsky score >70 (at initial cohort inclusion)
* Age ≥18 years old (at initial cohort inclusion)
* Completed follow-up in at least one previous study phase of the French HIV-HBV Cohort
* Obtained signed written informed consent

Exclusion Criteria:

* Refusal to participate
* Any severe physical, clinical or mental condition preventing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients with chronic hepatitis B.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03-31 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
HBV DNA replication | 14 years
  Proportion of patients with detectable HBV DNA levels, as determined by a commercially-available PCR assay (>60 international units/mL), at the beginning and end of follow-up
HBeAg-seroclearance | 14 years
  Proportion of hepatitis B "e" antigen (HBeAg)-positive patients who lose HBeAg-positive serology, as determined by a commercially-available ELISA assay, by the end of follow-up
HBsAg-seroclearance | 14 years
  Proportion of patients who lose hepatitis B surface antigen (HBsAg)-positive serology, as determined by a commercially-available ELISA assay, by the end of follow-up
Liver fibrosis (FibroTest) | 14 years
  Proportion of patients with equivalent F3 or F4 liver fibrosis, as determined by the FibroTest (non-invasive biochemical score) with a level >= 0.59, at the beginning and end of follow-up
Liver fibrosis (FibroScan) | 14 years
  Proportion of patients with equivalent F3 or F4 liver fibrosis, as determined by the FibroScan (transient elastography) with a level >= 7.6 kPa, at the beginning and end of follow-up

SECONDARY OUTCOMES:
Liver-related morbidity | 14 years
  Proportion of patients exhibiting any causes of morbidity related to liver-specific disease by the end of follow-up
Liver-related mortality | 14 years
  Proportion of patients who died due to liver-specific disease by the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boyd, MPH, PhD, Principal Investigator — INSERM UMR S 1136; Karine Lacombe, MD, PhD, Principal Investigator — INSERM UMR S 1136
Locations (4):
- France (4):
  - Centre hospitalier universitaire de Lyon, Lyon
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: Yes
Data will only be made available upon official request, pending approval by the Scientific Committee.

REFERENCES:
- [Background] Boyd A, Gozlan J, Miailhes P, Lascoux-Combe C, Cam MS, Rougier H, Zoulim F, Girard PM, Lacombe K. Rates and determinants of hepatitis B 'e' antigen and hepatitis B surface antigen seroclearance during long-term follow-up of patients coinfected with HIV and hepatitis B virus. AIDS. 2015 Sep 24;29(15):1963-73. doi: 10.1097/QAD.0000000000000795. PMID 26153669
- [Background] Boyd A, Gozlan J, Maylin S, Delaugerre C, Peytavin G, Girard PM, Zoulim F, Lacombe K. Persistent viremia in human immunodeficiency virus/hepatitis B coinfected patients undergoing long-term tenofovir: virological and clinical implications. Hepatology. 2014 Aug;60(2):497-507. doi: 10.1002/hep.27182. Epub 2014 Jun 20. PMID 24752996
- [Background] Lacombe K, Massari V, Girard PM, Serfaty L, Gozlan J, Pialoux G, Mialhes P, Molina JM, Lascoux-Combe C, Wendum D, Carrat F, Zoulim F. Major role of hepatitis B genotypes in liver fibrosis during coinfection with HIV. AIDS. 2006 Feb 14;20(3):419-27. doi: 10.1097/01.aids.0000200537.86984.0e. PMID 16439876